CLINICAL TRIAL: NCT00135954
Title: Treatment of Patients With Idiopathic Membranous Nephropathy at Risk for Renal Insufficiency: Comparison of Early Versus Late Start of Immunosuppressive Therapy
Brief Title: Treatment of Patients With Idiopathic Membranous Nephropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RUNMN01
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2007-02

CONDITIONS: Glomerulonephritis, Membranous
Keywords: membranous nephropathy; cyclophosphamide; prednisone
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Cyclophosphamide; Steroids; Prednisolone

ARMS (2):
- late intervention (Other): cyclophosphamide and steroids started at time of renal insufficiency
  Interventions: Drug: Cyclophosphamide and steroids
- early intervention (Experimental): immediate start of cyclophosphamide and steroids
  Interventions: Drug: Cyclophosphamide and steroids

INTERVENTIONS:
Drug: Cyclophosphamide and steroids — comparison of difference in time of start of therapy
  Other Names: prednisolone; endoxan

SUMMARY:
Patients with idiopathic membranous nephropathy at risk for renal failure can be identified in an early stage by measuring urinary low molecular weight proteins and urinary immunoglobulin G (IgG). This study evaluates the possible benefit of early start of immunosuppressive therapy in these high-risk patients.

DETAILED DESCRIPTION:
Inclusion Criteria:

* patients with idiopathic membranous nephropathy
* nephrotic syndrome
* normal renal function (serum creatinine [Screat] < 1.5 mg/dl)
* elevated urinary beta2-microglobulin and IgG

Immunosuppressive therapy consisting of:

* cyclophosphamide 1.5 mg/kg/day for 12 months
* prednisone orally, 0.5 mg/kg on alternate days for 6 months
* i.v. methylprednisolone 1000 mg on days 1,2,3, 60,61,62, 120,121,122

Study Groups:

* early: immediate start of immunosuppressive therapy at the time patient is identified as high-risk
* late: start of therapy after deterioration of renal function (increase of Screat > 25% and Screat > 1.5 mg/dl)

Main Outcome Parameters:

* serum creatinine
* remission of proteinuria
* period of nephrotic proteinuria
* major side effects: hospitalisations, infections

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic membranous nephropathy
* Serum creatinine < 1.5 mg/dl
* Nephrotic syndrome

Exclusion Criteria:

* Infection
* Instable angina
* Systemic disease
* Pregnancy
* Renal vein thrombosis
* Prior therapy with immunosuppressant agents
* Liver dysfunction
* Use of nonsteroidal anti-inflammatory drugs (NSAIDs)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 1997-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
renal function (serum creatinine)
proteinuria
side effects

CONTACTS AND LOCATIONS:
Overall Officials: Jack F Wetzels, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Department of Nephrology Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952
- [Derived] Hofstra JM, Branten AJ, Wirtz JJ, Noordzij TC, du Buf-Vereijken PW, Wetzels JF. Early versus late start of immunosuppressive therapy in idiopathic membranous nephropathy: a randomized controlled trial. Nephrol Dial Transplant. 2010 Jan;25(1):129-36. doi: 10.1093/ndt/gfp390. Epub 2009 Aug 8. PMID 19666912